CLINICAL TRIAL: NCT04049721
Title: Use of Hyperbaric Oxygen Therapy for the Treatment of Crush Injuries
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of manpower; logistic issues regarding the move of the in-hospital hyperbaric oxygen (HBO) chamber to an off-site location.
Sponsor: NYU Langone Health (Other)
Collaborators: Winthrop University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: s19-01074
Record Dates: First submitted 2019-07-30; First posted 2019-08-08 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Crush Injury
MeSH Terms: conditions — Crush Injuries | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care without HBO (Active Comparator): Intravenous access and fluid resuscitation (standard of care treatment)
  Interventions: Other: Standard of Care
- HBO + Standard of Care (Experimental): Ten daily treatment sessions of HBO at 2.5 atmospheres absolute (ATA) with 90 minutes of hyperbaric oxygen will be given over the course of two weeks
  Interventions: Procedure: HBO; Other: Standard of Care

INTERVENTIONS:
Procedure: HBO — 2.5 atmospheres absolute (ATA) with 90 minutes of hyperbaric oxygen will be given over the course of two weeks.
  Arms: HBO + Standard of Care
Other: Standard of Care — 20 patients will be included in the retrospective review arm. The retrospective chart review will be performed to determine the outcomes of patients with crush injuries treated at NYU Winthrop Hospital without HBO from 1/1/2012-12/31/2018.

SUMMARY:
The purpose of this study is to determine whether using hyperbaric oxygen (HBO) improves wound healing for patients who have a crush injury. The comparison of the prospective intervention group to the retrospective matched cohort aims to show that HBO can improve wound healing and decrease poor outcomes for patients with crush injuries. The information gained from this small study will serve as a basis for a follow-up prospective, randomized control trial to further delineate the role of HBO in a larger patient population.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to NYU Winthrop Hospital with a crush injury of the extremity, including appendages, up to 14 days post injury.
* No contraindication to hyperbaric oxygen therapy.
* Able and willing to sign informed consent.

Exclusion Criteria:

* Critically-ill patient requiring intubation or pressor support.
* Crush injury isolated to the distal phalanx (Tuft fracture).
* Absolute contraindication to hyperbaric oxygen therapy (untreated pneumothorax). Relative contraindications (uncontrolled congestive heart failure, uncontrolled seizure disorder, pulmonary disease, claustrophobia) will be assessed by the treating physician.
* Unable or unwilling to sign informed consent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
healing measured by percentage of skin necrosis using a Bilateral Perfusion Index (BPI; TCOM of the affected limb/TCOM of the nonaffected limb). | week 2
healing measured by percentage of skin necrosis using a Bilateral Perfusion Index (BPI; TCOM of the affected limb/TCOM of the nonaffected limb). | week 6
healing measured by percentage of skin necrosis using a Bilateral Perfusion Index (BPI; TCOM of the affected limb/TCOM of the nonaffected limb). | week 24
healing measured by percentage of skin necrosis using a Bilateral Perfusion Index (BPI; TCOM of the affected limb/TCOM of the nonaffected limb). | week 52

SECONDARY OUTCOMES:
hospital length of stay | 52 Weeks
  Number of days admitted over 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patrizio Petrone, MD, Principal Investigator — New York Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research
Access Criteria: The investigator who proposed to use the data.